CLINICAL TRIAL: NCT04384575
Title: Study on the Effectiveness of Gastroscope Operation Quality Control Based on Artificial Intelligence Technology
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Peng Yuan, MD,PHD, Peking University
Other Study IDs: PX2020047
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; artificial intelligence; endoscopy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Diagnostic Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blind spots — missed part during map the entire stomach through endoscopy

SUMMARY:
This study aims to construct a real-time quality monitoring system based on artificial intelligence technology.

DETAILED DESCRIPTION:
Gastroscopy plays an important role in the detection and diagnosis of upper gastrointestinal diseases. It is necessary for endoscopists to operate gastroscope according to the standardized process, in order to avoid missing early lesions. However, with the rapid increase in the number of endoscopies, the workload of endoscopists increases further. High workload reduces the quality of endoscopy, resulting in incomplete observation of anatomical parts that are easy to be missed in the process of gastroscopy. There are significant differences in the operation level of different endoscopists. Therefore, carrying out artificial intelligence methods has good academic research and practical value for improving the quality of endoscopic diagnosis and treatment.

Artificial intelligence devices need to use a large number of endoscopic images, based on this, we intends to collect endoscopic image data from our hospitals for training and validation of the model.

ELIGIBILITY:
Inclusion Criteria:

1. Patiens aged 18 years or above undergoing gastroscopy；
2. Be able to read, understand and sign informed consent；

Exclusion Criteria:

1. Patients with absolute contraindications to endoscopy examination;
2. pregnant women;
3. previous history of gastric surgery;
4. the researcher considers that the subject is not suitable for clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet the criteria for gastroscopy examination.
Sampling Method: Non-Probability Sample
Enrollment: 1570 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Accuracy | 2020.2.22-2020.7.1
  Calculate the accuracy of AI's judgment on images
Sensitivity | 2020.2.22-2020.7.1
  number of images in which AI correctly diagnosed positive/all images with positive
Specificity | 2020.2.22-2020.7.1
  number of images in which AI correctly diagnosed negative/all images negative

CONTACTS AND LOCATIONS:
Overall Officials: Qi Wu, MD., Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Haidian, China

REFERENCES:
- [Derived] Yuan P, Ma ZH, Yan Y, Li SJ, Wang J, Wu Q. Artificial Intelligence-Based Classification of Anatomical Sites in Esophagogastroduodenoscopy Images. Int J Gen Med. 2024 Dec 12;17:6127-6138. doi: 10.2147/IJGM.S481127. eCollection 2024. PMID 39691834